CLINICAL TRIAL: NCT02152085
Title: Neuromuscular Electrical Stimulation and Mobility in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Roger Enoka, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0720; R03HD079508 (NIH)
Record Dates: First submitted 2014-05-16; First posted 2014-06-02 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis
Keywords: Walking; Mobility; Neuromuscular electrical stimulation; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow pulse (Experimental): Six-week treatment of electrical stimulation applied to the calf muscles with stimulus pulses that last 0.4 ms.
  Interventions: Device: Narrow pulse
- Wide pulse (Experimental): Six-week treatment of electrical stimulation applied to the calf muscles with stimulus pulses that last 1 ms.
  Interventions: Device: Wide pulse

INTERVENTIONS:
Device: Narrow pulse — Participants will be randomly assigned to one of two study arms to receive a 6 week treatment of electrical stimulation that comprises narrow (0.4 ms) stimulus pulses.
  Arms: Narrow pulse
Device: Wide pulse — Participants will be randomly assigned to one of two study arms to receive a 6 week treatment of electrical stimulation that comprises wide (1 ms) stimulus pulses.
  Arms: Wide pulse

SUMMARY:
The purpose of this study is to investigate the capacity of a 6-week treatment with neuromuscular electrical stimulation to improve walking in individuals whose mobility has been compromised by multiple sclerosis.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two study arms. Those in one arm will receive a treatment with narrow stimulus pulses (0.4 ms) and those in the other arm will receive wide stimulus pulses (1 ms). The electrical stimulation will be delivered with a Vectra Genisys System.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and speak English to ensure safe participation in the project
* Difficulties with walking
* On stable doses of Ampyra, provigil, or other symptomatic-treating medications
* No systemic steroids within the last 30 days
* Not currently exercising more than 2x/wk
* Able to arrange own transportation to and from the laboratories
* Provide informed consent, including willingness to be randomly assigned to one of the two groups

Exclusion Criteria:

* Documented MS-related relapse in the last 3 months
* Medical diagnosis or condition that is considered to be an absolute or relative contraindication to participating in exercise training, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than treated basal cell cancer), other neurological disorders, or pregnancy
* Poorly controlled diabetes mellitus or hypertension
* History of seizure disorders
* Alcohol dependence or abuse (≥2 drinks/day), or present history (last 6 months) of drug abuse
* Inability to attend exercise sessions 3 days per week for 6 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Enoka, PhD, Principal Investigator — University of Colorado, Boulder; Jeffrey Hebert, PhD, PT, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three potential participants did not meet eligibility requirements.
Period: Overall Study
Arm/Group | Narrow Pulse | Wide Pulse
Started | 14 | 15
Completed | 13 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow Pulse | Wide Pulse | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9) | 55 (5) | 55 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Walking Endurance
Description: Distance walked in 6 min
Time Frame: Change from before to after 18 treatment sessions administered over a 6-week period (3 sessions/week).
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Narrow Pulse | Wide Pulse
Number analyzed (Participants) | 14 | 13
meters | 42 (60) | 25 (35)

2. Primary Outcome: Modified Fatigue Impact Scale
Description: MFIS scores range from 0 to 84 and higher numbers indicating worse fatigue.
Time Frame: Change from before to after 18 treatment sessions administered over a 6-week period (3 sessions/week).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Narrow Pulse | Wide Pulse
Number analyzed (Participants) | 14 | 13
score on a scale | 34 (17) | 23 (14)

3. Secondary Outcome: Maximal Walking Speed
Description: The time it takes to walk 25 ft
Time Frame: Change from before to after 18 treatment sessions administered over a 6-week period (3 sessions/week).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Narrow Pulse | Wide Pulse
Number analyzed (Participants) | 14 | 13
seconds | -1.92 (4.21) | 0.12 (1.15)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Narrow Pulse | Wide Pulse
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT02152085/Prot_000.pdf